CLINICAL TRIAL: NCT02064946
Title: High-dose Vitamin D Supplementation for ADT-induced Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Luke Peppone, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1R21CA175793-01A1 (NIH)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Neoplasms; Bone Mineral Density Quantitative Trait Locus 3
Keywords: prostate cancer; bone density; vitamin D; micronutrients; pharmacologic actions
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): Vitamin D3 50,000 IU: Patients will be assigned to receive weekly high-dose vitamin D (50,000 IU/week) along with a daily multivitamin (600 IU/day vitamin D + 210 mg/day calcium) and calcium supplements (1,000 mg/day calcium) for a period of 24 weeks.
  Interventions: Dietary Supplement: vitamin D
- Control (Placebo Comparator): Control: Patients will be assigned to receive a weekly vitamin D placebo along with a daily multivitamin (600 IU/day vitamin D + 210 mg/day calcium)and calcium supplements (1,000 mg/day calcium) for a period of 24 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — 50,000IU/week of vitamin D3
  Arms: Vitamin D3
Dietary Supplement: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to test the efficacy of a high-dose vitamin D supplementation regimen in reducing androgen deprivation therapy (ADT)-related side effects in older prostate cancer patients on ADT. The proposed study is a randomized, double-blind, 2-arm, controlled clinical trial that will accrue 76 prostate cancer patients without severe bone loss, aged 60 and older, beginning ADT, and scheduled to receive at least 6 months more of ADT. Participants will be randomized to: 1) weekly high-dose vitamin D3 (50,000 IU) or 2) vitamin D placebo only for a period of 24 weeks. Both groups will also receive a daily multivitamin and calcium supplement.

DETAILED DESCRIPTION:
The investigators hypothesize high-dose vitamin D supplementation will reduce androgen deprivation therapy (ADT)-related side effects including ADT-induced bone loss, decreased muscle mass, falls, reduced muscle strength, and diminished physical performance in older prostate cancer patients. The vitamin D supplementation is aimed at reducing fracture risk by maintaining proper bone density, thereby preventing osteoporotic/osteopenic conditions and increasing muscle mass. Both vitamin D and exercise are efficacious in maintaining proper bone health and muscle mass among the general population, but little research has been done on prostate cancer patients and survivors. Vitamin D could reduce fracture risk among prostate cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of stage I-IIIA prostate cancer
* Within 6 months of starting ADT with an additional 6 more months planned.
* Participants must have sub-optimal vitamin D levels of <32 ng/ml.
* Participants must agree not to take calcium and/or vitamin D supplements for the duration of the intervention other than those provided.
* Participants must have an ionized serum calcium level within normal limits (1.19-1.29mmol/L) and a total corrected serum calcium of ≤10.5 mg/dl.
* No contraindications for fitness testing and no physical limitations (e.g. cardiorespiratory, orthopedic, nervous system) as assessed by their physician.
* Able to read English (since the assessment materials are in printed format).
* Able to swallow medication and provide written informed consent.
* 60 years of age or older.

Exclusion Criteria:

* Previously verified diagnosis of osteoporosis (any t-score ≤ -2.5).
* Patients on antiresorptive drugs (i.e. bisphosphonates) within the past year.
* Patients with hypercalcemia (corrected serum Ca > 10.5 mg/dl) or a history of hypercalcemia or vitamin D toxicity/sensitivity.
* Patients with impaired renal function (CrCl < 60 mL/min) or who had kidney stones (calcium salt) within the past 5 years.
* Myocardial infarction within the past year.

Ages: 60 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
bone mineral density | after 24 weeks
  mean difference in bone mineral density between treatment group and control group
bone biomarkers | after 24 weeks
  amino-terminal collagen crosslinks (NTx) and bone-specific alkaline phosphatase (BSAP)

SECONDARY OUTCOMES:
muscle mass | after 24 weeks
  muscle mass as assessed by dual energy x-ray absorptiometry
muscular strength | after 24 weeks
  as assessed by Handgrip Dynamometer and 7-10 Repetition Maximum
physical performance | after 24 weeks
  as assessed by falls, physical performance battery, and 6-min walk test

CONTACTS AND LOCATIONS:
Overall Officials: Luke J Peppone, PhD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Wilmot Cancer Center, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Inglis JE, Fernandez ID, van Wijngaarden E, Culakova E, Reschke JE, Kleckner AS, Lin PJ, Mustian KM, Peppone LJ. Effects of High-Dose Vitamin D Supplementation on Phase Angle and Physical Function in Patients with Prostate Cancer on ADT. Nutr Cancer. 2021;73(10):1882-1889. doi: 10.1080/01635581.2020.1819348. Epub 2020 Sep 11. PMID 32911988